CLINICAL TRIAL: NCT05600205
Title: Evaluation of the Implementation and Effectiveness of a Combined Support for the Ambulatory Lifestyle Intervention (GOAL!)
Brief Title: Evaluation of Combined Support for the Ambulatory Lifestyle Intervention
Acronym: GOAL!
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: GGZ Centraal (Other)
Collaborators: ZonMw: The Netherlands Organisation for Health Research and Development (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 220307
Record Dates: First submitted 2022-10-26; First posted 2022-10-31 (Actual); Last update posted 2022-11-02 (Actual); Status verified 2022-10

CONDITIONS: Severe Mental Illness; Lifestyle
Keywords: Ambulatory; Implementation; Effectiveness
MeSH Terms: conditions — Mental Disorders

STUDY DESIGN:
Intervention Model Description: Quasi-experimental with a mixed-method matched design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- GOAL! (Experimental): Combined Support for the Ambulatory Lifestyle Intervention
  Interventions: Behavioral: GOAL!
- Control group (No Intervention): Care and counseling as usual (matched for gender, age and diagnosis)

INTERVENTIONS:
Behavioral: GOAL! — GOAL! is a integrated support focused on a combination of lifestyle factors for achieving a healthier lifestyle for people with severe mental illness. The intervention consists of two year of guidance from a lifestyle coach and qualified professionals.
  Arms: GOAL!

SUMMARY:
For people with a severe mental illness (SMI) there is no appropriate lifestyle intervention in ambulatory care, while they would benefit greatly from it. With SMI is meant mainly psychotic-, bipolar- and severe mood or anxiety disorders that require long-term care and counseling. People with SMI have a one-and-a-half to two times higher risk of heart disease, diabetes, and reduced mental health than the general population. This combination contributes to up to 15 years shorter life expectancy and reduced quality of life. Lifestyle plays an important role in this. Combined Support for the Ambulatory Lifestyle Intervention (GOAL!) is a multidisciplinary lifestyle support intervention where people with SMI are supervised for a longer period of time by qualified professionals, with attention to individual wishes and perceived challenges. Although the newly introduced so-called combined lifestyle interventions, that were recently introduced on a national level, follow this line of thinking, people with SMI may not benefit sufficiently from this offer. From the common challenge and need to create improved support, GGz Centraal in cooperation with the municipalities in the North Veluwe and local partners developed GOAL! and will pilot its use. This is done in cooperation with health insurers within the framework of an Innovation Policy Rule of the Dutch Healthcare Authority. The aim of this study is to follow this innovation and evaluate the implementation and effectiveness of GOAL!.

DETAILED DESCRIPTION:
Study design and setting

GOAL! will be evaluated through a quasi-experimental study with a mixed-method matched design. People with severe mental illness (SMI) receiving ambulatory care within the municipalities of North Veluwe will participate in the intervention. People who participate in GOAL! will be invited to additionally participate in its evaluation on a voluntary basis. Participants will be compared with a group of people with SMI who continue to receive usual counseling and care. This comparison group will be recruited outside municipalities where GOAL! takes place to avoid contamination. The aim is to recruit 50 participants of GOAL! for the evaluation and to create an equal comparison group of 50 participants matched for gender, age, and diagnosis. To evaluate the effects of GOAL! measurements will be conducted at baseline (T0), after 3 months (T1), after 12 months (T2), and after 24 months (T3).

Intervention

GOAL! aims to provide integrated support focused on a combination of lifestyle factors for achieving a healthier lifestyle for people with SMI. The intervention consists of one year of active guidance by the lifestyle coach, after which a maintenance program for another year is available. The participant starts with an intake interview with the lifestyle coach and then starts a basic course of three months in which participants have three group meetings of one hour each week. The group meetings focus on exercise (twice a week) and nutrition (once a week), and are given by qualified professionals in this field. After the basic course of three months a follow-up course of nine months starts with two group meetings of one hour per month given by the lifestyle coach. After the guidance phase of twelve months there is a maintenance program of also twelve months. This program consists of five sessions with individual counseling and three group meetings by the lifestyle coach.

Analysis

To measure the intervention effect, linear mixed models will be used. Although intervention and control groups are matched, potential differences between the groups on participant and disease characteristics are analyzed with independent t-tests (continuous variables) and chi-square tests (categorical variables). All models will be corrected for the baseline value, baseline disease severity, and monthly income category as a potential confounder for lifestyle behaviors. Corrections are made for potential clustering at the level of treatment team, neighborhood and municipality.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older;
* Diagnosed with a severe mental illness (SMI; defined as within treatment of a FACT team);
* Excessive abdominal circumference (≥102 cm for men or ≥ 88 cm for women; this is one of five risk factors for metabolic syndrome);
* Presence of at least one of the other four risk factors as clustered in the criteria for metabolic syndrome (hypertension, abnormal triglycerides, fasting blood sugar and HDL cholesterol, or medication use for blood pressure or values).

Exclusion Criteria:

* If someone lacks the legal capacity to give independent consent for participation and no (legal) representative is willing to give consent;
* If the disease severity at that time does not permit participation (i.e. acute psychological state, acute psychosis, or suicidality).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2022-11-01 (Estimated); Primary Completion 2025-11-01 (Estimated); Study Completion 2025-11-01 (Estimated)

PRIMARY OUTCOMES:
Change in physical activity: SIMPAQ | At baseline (T0), after 3 months (T1), after 12 months (T2) and after 24 months (T3)
  Measured by the Simple Physical activity Questionnaire (SIMPAQ). The SIMPAQ consists of five items (boxes), and participants are asked about time spent in bed (box 1), time sedentary, including naps (box 2), time spent walking (box 3), time spent exercising (box 4) and time spent in incidental activity, such as housekeeping (box 5). The total self-reported time spent on moderate-vigorous physical activity (MVPA) can be calculated by adding box 4 and 5.

SECONDARY OUTCOMES:
Change in dietary intake: MijnEetmeter | At baseline (T0), after 3 months (T1), after 12 months (T2) and after 24 months (T3)
  Measured by MijnEetmeter (dutch application) - a food diary. The participant fills in the nutritional intake for a given day. It provides insight into quantities of certain nutrients (i.e. fat, salt and sugar) and to what extent the participant ate according to the Schijf van Vijf (guideline for a healthy diet in the Netherlands) on that given day.
Change in sleep: SCOPA-SLEEP | At baseline (T0), after 3 months (T1), after 12 months (T2) and after 24 months (T3)
  Measured by the Scales for Outcomes in Parkinson's Disease - Sleep (SCOPA-Sleep). The SCOPA-Sleep is developed to evaluate night-time sleep and daytime sleepiness in a short and practical manner. The questionnaire enquires about the use of sleep medication and if so, which medication. It then uses 5 items to evaluate night-time sleep, 1 question inquiring overall quality of sleep followed by 6 items to evaluate daytime sleepiness on a 4 point Likert scale ranging from 0 (not at all) to 4 (a lot).
Change in substance use: ASSIST-Lite | At baseline (T0), after 3 months (T1), after 12 months (T2) and after 24 months (T3)
  The Alcohol, Smoking and Substance Involvement Screening Tool - Lite (ASSIST-Lite). Questions are about use, frequency, urges, health problems, control and concerns about various substances (including alcohol, opioids and soft drugs). Likert scales (Never, once or twice in my lifetime, monthly, weekly or daily; 0-4), and ordinal scales (Never; Yes, but not in the last three months; or Yes, but not in the last three months; scored 0,1,2) are used.
Change in weight | At baseline (T0), after 3 months (T1), after 12 months (T2) and after 24 months (T3)
  Weight is measured to the nearest 0.1 kg.
Change in BMI | At baseline (T0), after 3 months (T1), after 12 months (T2) and after 24 months (T3)
  Weight divided by height in meters squared
Change in metabolic health: waist circumference | At baseline (T0), after 3 months (T1), after 12 months (T2) and after 24 months (T3)
  Waist circumference measured halfway between the iliac crest and lowest rib in standing position
Change in metabolic health: systolic and diastolic blood pressure | At baseline (T0), after 3 months (T1), after 12 months (T2) and after 24 months (T3)
  Measured systolic and diastolic blood pressure (mmHg)
Change in fat percentage | At baseline (T0), after 3 months (T1), after 12 months (T2) and after 24 months (T3)
  Measured by the intelligent weighing scale, as the amount of body fat in relation to body weight (percentage on a scale from 0 to 100). A healthy fat percentage for men is between 7% to 25% and for women between 21% to 36%. Fat percentage increases with age.
Change in psychopathology: BSI | At baseline (T0), after 3 months (T1), after 12 months (T2) and after 24 months (T3)
  Measured by the Brief Symptom Inventory (BSI). The BSI comprises 53 items that reflect 9 symptom domains of psychopathology (somatization, obsessive compulsive, interpersonal sensitivity, depression, anxiety, hostility, phobic anxiety, paranoid ideation and psychoticism). Each item is rated on a 5-point scale of distress from 0 (not at all) to 4 (extremely).
Change in Quality of life: EQ-5D | At baseline (T0), after 3 months (T1), after 12 months (T2) and after 24 months (T3)
  Measured by the EuroQol 5D (EQ-5D).The EQ-5D is a generic instrument that consists of 5 dimensions of health, with one item per dimension; mobility, selfcare, usual activities, pain/discomfort, and anxiety/depression. There are three levels of severity ranging from no issues to many issues. The index score are calculated ranging from 0 (worst quality of life) to 1 (perfect quality of life).
Change care use and illness and work: TIC-P | At baseline (T0) and after 24 months (T3)
  De Treatment Inventory of Costs in Patients with psychiatric disorders (TiC-P). Dutch questionnaire for the evaluation of costs related to psychosocial problems, consisting of three parts.15 questions are about certain facilities in (mental) health care (part 1), 11 questions are about the extent to which psychosocial problems hindered the respondent in (paid and unpaid) work (part 2) and part three consists of some general questions. To arrive at a total cost score, the frequency of care consumption/productivity loss is multiplied by the related costs according to national guidelines.
Barriers and facilitators of the implementation of GOAL!: MIDI | At baseline (T0) and after 24 months (T3)
  Measured by the Measurement Instrument for Determinants of the Innovation (MIDI). The MIDI is comprised of 28 items, divided into 4 scales measuring determinants associated with innovations (7 items), the user (11 items) and the organization (10 items). All items are scored on a 5-point Likert scale ranging from 1 (totally disagree) to 5 (totally agree). Items which ≥20% responds negatively (disagree/totally disagree) are considered barriers. Items which ≥80% respond positively (agree/totally agree) are considered facilitators.

OTHER OUTCOMES:
Achieving lifestyle goals | 24 months
  Questioned and reported by the lifestyle coach on an ongoing basis.
Adverse events | 24 months
  Evaluated by the lifestyle coach on an ongoing basis.

CONTACTS AND LOCATIONS:
Locations (1):
- GGz Centraal, Amersfoort, Utrecht, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hjorthoj C, Sturup AE, McGrath JJ, Nordentoft M. Years of potential life lost and life expectancy in schizophrenia: a systematic review and meta-analysis. Lancet Psychiatry. 2017 Apr;4(4):295-301. doi: 10.1016/S2215-0366(17)30078-0. Epub 2017 Feb 22. PMID 28237639
- [Background] Correll CU, Solmi M, Veronese N, Bortolato B, Rosson S, Santonastaso P, Thapa-Chhetri N, Fornaro M, Gallicchio D, Collantoni E, Pigato G, Favaro A, Monaco F, Kohler C, Vancampfort D, Ward PB, Gaughran F, Carvalho AF, Stubbs B. Prevalence, incidence and mortality from cardiovascular disease in patients with pooled and specific severe mental illness: a large-scale meta-analysis of 3,211,768 patients and 113,383,368 controls. World Psychiatry. 2017 Jun;16(2):163-180. doi: 10.1002/wps.20420. PMID 28498599
- [Background] Deenik J, Czosnek L, Teasdale SB, Stubbs B, Firth J, Schuch FB, Tenback DE, van Harten PN, Tak ECPM, Lederman O, Ward PB, Hendriksen IJM, Vancampfort D, Rosenbaum S. From impact factors to real impact: translating evidence on lifestyle interventions into routine mental health care. Transl Behav Med. 2020 Oct 8;10(4):1070-1073. doi: 10.1093/tbm/ibz067. PMID 31169897
- [Background] Deenik J, Tenback DE, Tak ECPM, Hendriksen IJM, van Harten PN. [Thinking inside the box: improving the lifestyle of inpatients with severe mental illness]. Tijdschr Psychiatr. 2020;62(7):564-574. Dutch. PMID 32700302
- [Background] Firth J, Siddiqi N, Koyanagi A, Siskind D, Rosenbaum S, Galletly C, Allan S, Caneo C, Carney R, Carvalho AF, Chatterton ML, Correll CU, Curtis J, Gaughran F, Heald A, Hoare E, Jackson SE, Kisely S, Lovell K, Maj M, McGorry PD, Mihalopoulos C, Myles H, O'Donoghue B, Pillinger T, Sarris J, Schuch FB, Shiers D, Smith L, Solmi M, Suetani S, Taylor J, Teasdale SB, Thornicroft G, Torous J, Usherwood T, Vancampfort D, Veronese N, Ward PB, Yung AR, Killackey E, Stubbs B. The Lancet Psychiatry Commission: a blueprint for protecting physical health in people with mental illness. Lancet Psychiatry. 2019 Aug;6(8):675-712. doi: 10.1016/S2215-0366(19)30132-4. Epub 2019 Jul 16. No abstract available. PMID 31324560
- [Background] Firth J, Solmi M, Wootton RE, Vancampfort D, Schuch FB, Hoare E, Gilbody S, Torous J, Teasdale SB, Jackson SE, Smith L, Eaton M, Jacka FN, Veronese N, Marx W, Ashdown-Franks G, Siskind D, Sarris J, Rosenbaum S, Carvalho AF, Stubbs B. A meta-review of "lifestyle psychiatry": the role of exercise, smoking, diet and sleep in the prevention and treatment of mental disorders. World Psychiatry. 2020 Oct;19(3):360-380. doi: 10.1002/wps.20773. PMID 32931092
- [Background] Suetani S, Rosenbaum S, Scott JG, Curtis J, Ward PB. Bridging the gap: What have we done and what more can we do to reduce the burden of avoidable death in people with psychotic illness? Epidemiol Psychiatr Sci. 2016 Jun;25(3):205-10. doi: 10.1017/S2045796015001043. Epub 2016 Jan 15. PMID 26768358
- [Background] Firth J, Ward PB, Stubbs B. Editorial: Lifestyle Psychiatry. Front Psychiatry. 2019 Aug 26;10:597. doi: 10.3389/fpsyt.2019.00597. eCollection 2019. No abstract available. PMID 31507466
- [Derived] Noortman-van Meteren CR, van Schothorst MME, den Bleijker NM, Braakhuis-Keuning B, Houwert-Zuidema WMH, van Amelsvoort TAMJ, Deenik J. (Cost-)effectiveness and implementation of a combined lifestyle intervention for outpatients with severe mental illness (GOAL!): a hybrid quasi-experimental study protocol. BMC Psychiatry. 2024 Nov 14;24(1):804. doi: 10.1186/s12888-024-06216-x. PMID 39543515